CLINICAL TRIAL: NCT01126541
Title: A Comparative Study to Assess the Effect of Retreatment With 2 Doses of MabThera on Disease Activity Score in Patients With Active Rheumatoid Arthritis Who Have Had an Inadequate Response or Intolerance to antiTNF-alfa Therapy.(SMART)
Brief Title: SMART Study: A Study of Re-treatment With MabThera (Rituximab) in Patients With Rheumatoid Arthritis Who Have Failed on Anti-TNF Alfa Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML19895
Record Dates: First submitted 2010-05-18; First posted 2010-05-19 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

ARMS (2):
- A (Experimental): 1000 mg IV rituximab
  Interventions: Drug: rituximab
- B (Experimental): 2 x 1000 mg IV rituximab
  Interventions: Drug: rituximab

INTERVENTIONS:
Drug: rituximab — Arm A: 1000 mg IV (one infusion) every 2 months \nArm B: 2 x 1000 mg IV (2 infusions) every 2 months
  Other Names: MabThera/Rituxan

SUMMARY:
This study will compare the efficacy and safety of re-treatment with 2 doses of MabThera (rituximab) in patients with active rheumatoid arthritis (RA) who have previously experienced an inadequate response or intolerance to anti-tumor necrosis factor (anti-TNF) therapies etanercept, infliximab or adalimumab therapy. All patients will receive infusions of 1000 mg intravenous (IV) MabThera on Days 1 and 15; at Week 24 patients who have demonstrated a moderate or good response will be randomized to receive re-treatment with either 1 or 2 additional infusions of 1000 mg IV MabThera. The anticipated time on study treatment is 2+ years, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >18 years of age
* RA for >=6 months
* Receiving outpatient treatment
* Ongoing treatment with methotrexate for >=3 months, stable for >=1 month
* Inadequate response or intolerance to etanercept, infliximab or adalimumab

Exclusion Criteria:

* Previous treatment with MabThera
* Concurrent treatment with any anti TNF-alfa therapy or biologic therapy
* Previous treatment with any investigational cell-depleting therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2006-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (46):
- France (46):
  - Abbeville
  - Agen
  - Aix-en-Provence
  - Aix-les-Bains
  - Amiens
  - Belfort
  - Berck
  - Bobigny
  - Bois-Guillaume
  - Boulogne-Billancourt
  - Brest
  - Caen
  - Cahors
  - Clermont-Ferrand
  - Corbeil-Essonnes
  - Échirolles
  - La Roche-sur-Yon
  - Le Kremlin-Bicêtre
  - Libourne
  - Liévin
  - Lille
  - Limoges
  - Lomme
  - Lyon
  - Marseille
  - Montivilliers
  - Montpellier
  - Nantes
  - Narbonne
  - Nice
  - Paris
  - Pau
  - Perpignan
  - Pessac
  - Pierre-Bénite
  - Poitiers
  - Reims
  - Rennes
  - Saint-Etienne
  - Strasbourg
  - Toulon
  - Toulouse
  - Valence
  - Valenciennes
  - Vandœuvre-lès-Nancy
  - Vannes

REFERENCES:
- [Derived] de Jong TD, Sellam J, Agca R, Vosslamber S, Witte BI, Tsang-A-Sjoe M, Mantel E, Bijlsma JW, Voskuyl AE, Nurmohamed MT, Verweij CL, Mariette X. A multi-parameter response prediction model for rituximab in rheumatoid arthritis. Joint Bone Spine. 2018 Mar;85(2):219-226. doi: 10.1016/j.jbspin.2017.02.015. Epub 2017 Mar 28. PMID 28363827
- [Derived] Sellam J, Riviere E, Courties A, Rouzaire PO, Tolusso B, Vital EM, Emery P, Ferraccioli G, Soubrier M, Ly B, Hendel Chavez H, Taoufik Y, Dougados M, Mariette X. Serum IL-33, a new marker predicting response to rituximab in rheumatoid arthritis. Arthritis Res Ther. 2016 Dec 13;18(1):294. doi: 10.1186/s13075-016-1190-z. PMID 27964756
- [Derived] Sellam J, Rouanet S, Hendel-Chavez H, Miceli-Richard C, Combe B, Sibilia J, Le Loet X, Tebib J, Jourdan R, Dougados M, Taoufik Y, Mariette X. CCL19, a B cell chemokine, is related to the decrease of blood memory B cells and predicts the clinical response to rituximab in patients with rheumatoid arthritis. Arthritis Rheum. 2013 Sep;65(9):2253-61. doi: 10.1002/art.38023. PMID 23740460
- [Derived] Mariette X, Rouanet S, Sibilia J, Combe B, Le Loet X, Tebib J, Jourdan R, Dougados M. Evaluation of low-dose rituximab for the retreatment of patients with active rheumatoid arthritis: a non-inferiority randomised controlled trial. Ann Rheum Dis. 2014 Aug;73(8):1508-14. doi: 10.1136/annrheumdis-2013-203480. Epub 2013 May 30. PMID 23723317
- [Derived] Sellam J, Rouanet S, Hendel-Chavez H, Abbed K, Sibilia J, Tebib J, Le Loet X, Combe B, Dougados M, Mariette X, Taoufik Y. Blood memory B cells are disturbed and predict the response to rituximab in patients with rheumatoid arthritis. Arthritis Rheum. 2011 Dec;63(12):3692-701. doi: 10.1002/art.30599. PMID 22127692
- [Derived] Sellam J, Hendel-Chavez H, Rouanet S, Abbed K, Combe B, Le Loet X, Tebib J, Sibilia J, Taoufik Y, Dougados M, Mariette X. B cell activation biomarkers as predictive factors for the response to rituximab in rheumatoid arthritis: a six-month, national, multicenter, open-label study. Arthritis Rheum. 2011 Apr;63(4):933-8. doi: 10.1002/art.30233. PMID 21225699

RESULTS

PARTICIPANT FLOW:
Groups:
- Randomized Retreatment Arm A: Rituximab 1000 Milligrams (mg): Participants received rituximab 1000 mg intravenously (IV) on Days 1 and 15. After Week 24, if Disease Activity Score based on 28-Joint Count (DAS28) was greater than (>)3.2, participants received one additional infusion of rituximab 1000 mg IV. Participants received methylprednisolone 100 mg IV 30 minutes before each rituximab infusion and methotrexate (MTX) ≥10 milligrams per week (mg/week) by mouth or parenteral throughout course of treatment.
- Randomized Retreatment Arm B: Rituximab 1000 mg x 2: Participants received rituximab 1000 mg IV on Days 1 and 15. After Week 24, if DAS28 was >3.2, participants received two additional infusions of rituximab 1000 mg IV, 15 days apart. Participants received methylprednisolone 100 mg IV 30 minutes before each rituximab infusion and ≥10 mg/week MTX by mouth or parenteral throughout course of treatment.
- Nonrandomized: Rituximab 1000 mg: Participants received rituximab 1000 mg IV on Days 1 and 15, methylprednisolone 100 mg IV at 30 minutes before each rituximab infusion, and MTX ≥10 mg/week by mouth or parenterally throughout treatment course.
Period: Overall Study
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 Milligrams (mg) | Randomized Retreatment Arm B: Rituximab 1000 mg x 2 | Nonrandomized: Rituximab 1000 mg
Started | 70 | 73 | 81
Completed | 60 | 61 | 55
Not Completed | 10 | 12 | 26
Not completed — Adverse Event | 0 | 2 | 4
Not completed — Death | 0 | 1 | 0
Not completed — Lack of Efficacy | 6 | 1 | 11
Not completed — Lost to Follow-up | 1 | 2 | 2
Not completed — Withdrawal by Subject | 2 | 5 | 6
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Administrative reason or other | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Randomized Retreatment Arm A: Rituximab 1000 mg: Participants received rituximab 1000 mg IV on Days 1 and 15. After Week 24, if DAS28 was >3.2, participants received one additional infusion of rituximab 1000 mg IV. Participants received methylprednisolone 100 mg IV 30 minutes before each rituximab infusion and MTX ≥10 mg/week by mouth or parenteral throughout course of treatment.
- Total: Total of all reporting groups
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2 | Nonrandomized: Rituximab 1000 mg | Total
Number analyzed (Participants) | 70 | 73 | 81 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (11.5) | 57.2 (10.4) | 56.1 (11.2) | 56.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 62 | 70 | 187
  Male | 15 | 11 | 11 | 37

OUTCOME MEASURES:

1. Secondary Outcome: DAS28-CRP During the Initial Treatment
Description: Mean DAS28-CRP at Week 24 of the Initial Treatment study. DAS28-CRP was based on joint counts, overall participant assessment, and the serum CRP level at each visit. Joint counts included SJC and TJC using the 28 joints count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-CRP ≤3.2 implied low disease activity, >3.2 to 5.1 implied moderate to high disease activity, and <2.6=remission.
Time Frame: Days 1 and 15, and Weeks 6, 12, and 24
Population: Overall population: all participants with at least one treatment intake.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Randomized Group: Participants received rituximab 1000 mg IV on Days 1 and 15. After Week 24, if DAS28 was >3.2, participants were randomized to receive a single rituximab 1000 mg IV infusion (Retreatment Arm A) or 2 x rituximab 1000 mg IV infusions 15 days apart (Retreatment Arm B). All participants received methylprednisolone 100 mg IV 30 minutes before each rituximab infusion and MTX ≥10 mg/week by mouth or parenteral throughout course of treatment.
- Nonrandomized Group: Participants received rituximab 1000 mg IV on Days 1 and 15, methylprednisolone 100 mg IV at 30 minutes before each rituximab infusion, and MTX ≥10 mg/week by mouth or parenterally throughout treatment course.
Arm/Group | Randomized Group | Nonrandomized Group
Number analyzed (Participants) | 143 | 81
units on a scale
  First Course, Day 1 | 5.82 (0.85) | 5.77 (0.90)
  First Course, Day 15 | 5.33 (1.09) | 5.42 (1.07)
  Follow-up, Week 6 | 4.69 (0.95) | 5.12 (1.05)
  Follow-up, Week 12 | 4.13 (0.91) | 5.00 (1.19)
  Follow-up, Week 24 | 3.65 (0.85) | 5.24 (1.08)

2. Secondary Outcome: DAS28-CRP and Changes From Baseline to Week 24 in DAS28-CRP by Retreatment Course
Description: DAS28-CRP was based on joint counts, overall participant assessment, and the serum CRP level at each visit. Joint counts included SJC and TJC using the 28 joints count and CRP (mg/L). Total score range=0 to 9.4; a higher score indicated more disease activity. A DAS28-CRP score of ≤3.2 implied low disease activity, >3.2 to 5.1 implied moderate to high disease activity, and <2.6=remission.
Time Frame: Day 1, 24 weeks following each infusion up to 72 Weeks
Population: ITT Population; number (n)=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 70 | 73
units on a scale
  Initial treatment, Day 1 (n=70,73) | 5.79 (0.85) | 5.84 (0.86)
  Initial treatment, Week 24 (n=70,73) | 3.57 (0.89) | 3.73 (0.80)
  Change at Week 24 (n=70,73) | -2.22 (0.96) | -2.11 (0.93)
  1st retreatment, Day 1 (n=66,68) | 4.33 (0.91) | 4.45 (0.80)
  1st retreatment, Week 24 (n=66,68) | 3.67 (1.15) | 3.69 (1.05)
  1st retreatment, Change at Week 24 (n=66,68) | -0.67 (1.15) | -0.79 (1.13)
  2nd retreatment, Day 1 (n=49,48) | 4.60 (0.87) | 4.55 (0.96)
  2nd retreatment, Week 24 (n=41,39) | 3.72 (1.10) | 3.76 (1.12)
  2nd retreatment, Change at Week 24 (n=41,39) | -0.94 (1.17) | -0.78 (1.07)
Statistical Analysis 1: Comparison: Randomized Retreatment Arm A: Rituximab 1000 mg vs Randomized Retreatment Arm B: Rituximab 1000 mg x 2; Change from Day 1 to Week 24 (initial treatment); Test type: Non-Inferiority or Equivalence — Primary objective to demonstrate noninferiority of retreatment with one 1000 mg rituximab infusion. Mean ±SD of the DAS28-CRP AUC at 24 months = 2218 ±967 (based on EDWARDS, REFLEX and DANCER study data). H0 (null hypothesis): Arm B - Arm A >20%. H1: Arm B - Arm A ≤ 20%. Power = 80%; Larger difference clinically acceptable = 20% = 444; Significance level of 2.5% (one-sided); p = 0.465, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Randomized Retreatment Arm A: Rituximab 1000 mg vs Randomized Retreatment Arm B: Rituximab 1000 mg x 2; Arm A vs. Arm B: Change from 1st retreatment to 24 weeks after; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.161, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Randomized Retreatment Arm A: Rituximab 1000 mg vs Randomized Retreatment Arm B: Rituximab 1000 mg x 2; Arm A vs. Arm B: Change from 2nd retreatment to 24 weeks after; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.524, Student t-test

3. Primary Outcome: Disease Activity Score Based on 28-Joints Count and C-Reactive Protein (DAS28-CRP) Area Under the Curve (AUC) at Week 104
Description: DAS28-CRP was based on joint counts, overall participant assessment, and serum CRP levels (measured in milligrams per liter [mg/L]) at each visit. Joint counts included swollen joint count (SJC) and tender joint count (TJC). Total score range was 0 to 9.4; a higher score indicated more disease activity. DAS28-CRP less than or equal to (≤)3.2 implied low disease activity, >3.2 to 5.1 implied moderate to high disease activity, and less than (<)2.6 equals (=) remission. The AUC of all DAS28-CRP values between Day 1 and Week 104 (15 values of protocol visits) was calculated using the trapeze method (AUC between t1 and t2=(t2-t1)*((DAS28-CRP at t1 + DAS28-CRP at t2)/2). The true visit dates were used to calculate the time between 2 DAS28-CRP evaluations. All the AUC were censored at Week 104 (linear extrapolation using the 2 last DAS28-CRP values (Weeks 96 and 104) to obtain the "true" DAS28-CRP value at the "true" Week 104).
Time Frame: Week 104
Population: Per Protocol (PP) population: all randomized participants in the Intent-to-Treat (ITT) population (defined as all randomized participants) without major protocol violations. Participants were grouped according to their initially assigned treatment arm irrespective of the treatment actually received.
Measure: Mean (Standard Error); unit: score on a scale*week
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 51 | 49
score on a scale*week | 2761.4 (507.8) | 2666.0 (490.4)
Statistical Analysis 1: Comparison: Randomized Retreatment Arm A: Rituximab 1000 mg vs Randomized Retreatment Arm B: Rituximab 1000 mg x 2; Test type: Non-Inferiority or Equivalence — Primary objective to demonstrate noninferiority of retreatment with one 1000 mg rituximab infusion. Mean plus or minus (±)SD of the DAS28-CRP AUC at 24 months = 2218 ±967 (based on EDWARDS, REFLEX and DANCER study data). H0 (null hypothesis): Arm B - Arm A >20%. H1: Arm B - Arm A ≤ 20%. Power = 80%; Larger difference clinically acceptable = 20% = 444; Significance level of 2.5% (one-sided); Adjusted difference = 51.38, 95% CI 2-sided [-131.22 to 233.98], Standard Deviation 92.00 — Covariate analysis with baseline DAS28-CRP value as covariate

4. Secondary Outcome: Percentage of Participants Achieving Clinical Remission (DAS28-CRP <2.6) or Low Disease Activity (DAS28-CRP ≤3.2)
Description: Percentage of participants with clinical remission and low disease activity as measured by DAS28-CRP for Arm A and Arm B at Week 24 of the Initial Treatment, at 24 weeks after first re-treatment, and at 24 weeks after second retreatment. DAS28-CRP was based on joint counts, overall participant assessment, and the serum CRP level at each visit. Joint counts included SJC and TJC using the 28 joints count and CRP (mg/L). Total score range=0 to 9.4; a higher score indicated more disease activity. A DAS28-CRP score of ≤3.2 implied low disease activity and <2.6 = remission.
Time Frame: Week 24 of the Initial Treatment, 24 weeks after first retreatment, and 24 weeks after second retreatment
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 70 | 73
percentage of participants
  Remission: Initial Treatment, Week 24 (n=70,73) | 14.3 | 8.2
  Remission: 1st Re-treatment, Week 24 (n=66,67) | 18.2 | 9.0
  Remission: 2nd Retreatment, Week 24 (n=43,40) | 16.3 | 7.5
  Low activity: Initial Treatment, Week 24 (n=70,73) | 37.1 | 27.4
  Low activity: 1st Retreatment, Week 24 (n=66,67) | 34.8 | 35.8
  Low activity: 2nd Retreatment, Week 24 (n=43,40) | 27.9 | 30.0

5. Secondary Outcome: DAS28-CRP AUC Weighted Time
Description: as for outcome 2
Time Frame: Days 1 and 15, Weeks 6, 12, and 24 and every 8 weeks thereafter through Week 104
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale*week
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 70 | 73
units on a scale*week | 3.82 (0.71) | 3.88 (0.71)

6. Secondary Outcome: Time to Achieve DAS28-CRP Remission After the First Course
Description: DAS28-CRP was based on joint counts, overall participant assessment, and the serum CRP level at each visit. Joint counts included SJC and TJC using the 28 joints count and CRP (mg/L). Total score range=0 to 9.4; a higher score indicated more disease activity. A DAS28-CRP <2.6=remission.
Time Frame: Days 1 and 15, Weeks 6, 12, and 24 and every 8 weeks thereafter through Week 104
Population: ITT population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Randomized Group
Number analyzed (Participants) | 143
weeks | 56.0 [34.9 to NA] — Upper limit of the 95% confidence interval (CI) for the time to remission could not be calculated due to an insufficient number of events occurring.

7. Secondary Outcome: Time to Achieve DAS28-CRP Remission After Retreatment
Description: as for outcome 6
Time Frame: Days 1 and 15, Weeks 6, 12, and 24 and every 8 weeks thereafter through Week 104
Population: ITT population; n=number of participants assessed at a given visit.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 66 | 68
weeks
  1st retreatment (n=66,68) | NA [NA to NA] — Time to remission could not be determined due to an insufficient number of events occurring. | 78.1 [37.0 to NA] — Upper limit of the 95% CI for time to remission could not be determined due to an insufficient number of events occurring.
  2nd retreatment (n=49,48) | NA [NA to NA] — Time to remission could not be determined due to an insufficient number of events occurring. | NA [NA to NA] — Time to remission could not be determined due to an insufficient number of events occurring.

8. Secondary Outcome: Time to Achieve DAS28-CRP ≤3.2 After the First Course of Treatment
Description: DAS28-CRP was based on joint counts, overall participant assessment, and the serum CRP level at each visit. Joint counts included SJC and TJC using the 28 joints count and CRP (mg/L). Total score range=0 to 9.4; a higher score indicated more disease activity. A DAS28-CRP score of ≤3.2 implied low disease activity.
Time Frame: Days 1 and 15, Weeks 6, 12, and 24 and every 8 weeks thereafter through Week 104
Population: ITT population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Randomized Group
Number analyzed (Participants) | 143
weeks | 28.0 [25.4 to NA] — Upper limit of the 95% CI for time to low disease activity could not be calculated due to an insufficient number of events occurring.

9. Secondary Outcome: Time to Achieve DAS28-CRP ≤3.2 After Retreatment
Description: as for outcome 8
Time Frame: Days 1 and 15, Weeks 6, 12, and 24 and every 8 weeks thereafter through Week 104
Population: ITT population; n=number of participants assessed at a given visit.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 66 | 68
weeks
  1st retreatment (n=66,68) | 31.0 [21.1 to NA] — Upper limit of the 95% CI for time to low disease activity could not be calculated due to an insufficient number of events occurring. | 22.1 [14.1 to 47.9]
  2nd retreatment (n=49,48) | 16.9 [14.1 to 33.9] | 29.0 [15.0 to NA] — Upper limit of the 95% CI for time to low disease activity could not be calculated due to an insufficient number of events occurring.

10. Secondary Outcome: Duration of DAS28-CRP Remission After the First Course of Treatment
Description: as for outcome 6
Time Frame: Days 1 and 15, Weeks 6, 12, and 24 and every 8 weeks thereafter through Week 104
Population: ITT population; only participants with a response (DAS28-CRP <2.6) during initial treatment (at any point) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Randomized Group
Number analyzed (Participants) | 34
weeks | 11.7 [8.0 to 15.1]

11. Secondary Outcome: Duration of DAS28-CRP Remission After Retreatment
Description: as for outcome 6
Time Frame: Days 1 and 15, Weeks 6, 12, and 24 and every 8 weeks thereafter through Week 104
Population: ITT population; only participants with a response (DAS28-CRP <2.6) during retreatment (at any point) were included in the analysis. n=number of participants assessed at a given visit.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 21 | 22
weeks
  1st retreatment (n=21,22) | 16.0 [15.0 to 17.0] | 8.0 [7.7 to 15.1]
  2nd retreatment (n=17,11) | 9.0 [8.0 to 16.3] | 8.0 [8.0 to 16.0]

12. Secondary Outcome: Duration of DAS28-CRP ≤3.2 After the First Course of Treatment
Description: as for outcome 8
Time Frame: Days 1 and 15, Weeks 6, 12, and 24 and every 8 weeks thereafter through Week 104
Population: ITT population; only participants with a response (DAS28-CRP ≤3.2) during first course of treatment (at any point) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Randomized Group
Number analyzed (Participants) | 65
weeks | 14.3 [9.0 to 18.6]

13. Secondary Outcome: Duration of DAS28-CRP ≤3.2 After Retreatment
Description: as for outcome 8
Time Frame: Days 1 and 15, Weeks 6, 12, and 24 and every 8 weeks thereafter through Week 104
Population: ITT population; only participants with a response (DAS28-CRP ≤3.2) during retreatment (at any point) were included in the analysis. n=number of participants assessed at a given visit.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 35 | 40
weeks
  1st retreatment (n=35,40) | 27.0 [22.7 to 32.0] | 17.0 [9.0 to 28.0]
  2nd retreatment (n=29,23) | 10.1 [8.0 to 32.1] | 16.0 [9.0 to 31.1]

14. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20%, 50%, and 70% Improvement (ACR20/ACR50/ACR70)
Description: ACR20/50/70 response defined as ≥20%, 50%, or 70% improvement, respectively, in TJC and SJC, and ≥20%, 50%, or 70% improvement, respectively, in at least 3 of 5 remaining ACR core measures: Patient Global Assessment of Pain, Patient's Global Assessment of Disease Activity, Physician's Global Assessment of Disease Activity (on a visual analog scale [VAS]); Health Assessment Questionnaire-Disability Index (HAQ-DI); and CRP.
Time Frame: Week 24 of the initial treatment, 24 weeks after first retreatment, and 24 weeks after second retreatment
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 70 | 73
percentage of participants
  ACR20: Initial Treatment, Week 24 | 78.6 | 75.3
  ACR20: 1st Retreatment, Week 24 | 63.6 | 61.2
  ACR20: 2nd Retreatment, Week 24 | 65.1 | 60.0
  ACR50: Initial Treatment, Week 24 | 35.7 | 32.9
  ACR50: 1st Retreatment, Week 24 | 33.3 | 32.8
  ACR50: 2nd Retreatment, Week 24 | 32.6 | 42.5
  ACR70: Initial Treatment, Week 24 | 12.9 | 11.0
  ACR70: 1st Retreatment, Week 24 | 16.7 | 19.4
  ACR70: 2nd Retreatment, Week 24 | 18.6 | 20.0

15. Secondary Outcome: Percentage of Participants Achieving a Response During Initial Treatment by European League Against Rheumatism (EULAR) Category
Description: DAS28-based EULAR response criteria were used to measure individual response as no response, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders = change from baseline >1.2 with a DAS28 score of ≤3.2; moderate responders = change from baseline >1.2 with a DAS28 score of >3.2 to ≤ 5.1 or change from baseline >0.6 to ≤1.2 with a DAS28 score of ≤5.1; non-responders = change from baseline ≤0.6 or change from baseline >0.6 and ≤ 1.2 with a DAS28 score of >5.1.
Time Frame: Day 15, Weeks 6, 12, and 24
Population: Overall population
Measure: Number; unit: percentage of participants
Arm/Group | Randomized Group | Nonrandomized Group
Number analyzed (Participants) | 143 | 81
percentage of participants
  Good response: Day 15 | 4 | 3
  Good response: Week 6 | 5 | 4
  Good response: Week 12 | 15 | 4
  Good response: Week 24 | 32 | 3
  Moderate response: Day 15 | 22 | 20
  Moderate response: Week 6 | 59 | 29
  Moderate response: Week 12 | 73 | 35
  Moderate response: Week 24 | 66 | 15
  No response: Day 15 | 74 | 78
  No response: Week 6 | 36 | 67
  No response: Week 12 | 11 | 61
  No response: Week 24 | 3 | 82

16. Secondary Outcome: Percentage of Participants Achieving a Response During Retreatment by EULAR Category
Description: as for outcome 15
Time Frame: Week 24, 24 weeks after 1st retreatment, 24 weeks after 2nd retreatment
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 70 | 73
percentage of participants
  Good response: Week 24 (n=70,73) | 37 | 26
  Good response: 1st retreatment (n=66,67) | 35 | 36
  Good response: 2nd retreatment (n=43,40) | 28 | 30
  Moderate response: Week 24 (n=70,73) | 60 | 71
  Moderate response: 1st retreatment (n=66,67) | 53 | 52
  Moderate response: 2nd retreatment (n=43,40) | 54 | 50
  No response: Week 24 (n=70,73) | 3 | 3
  No response: 1st retreatment (n=66,67) | 12 | 12
  No response: 2nd retreatment (n=43,40) | 19 | 20

17. Secondary Outcome: Percentage of Participants With Rheumatoid Factor (RF) at 24 Weeks After Treatment
Description: RF is the auto antibody directed against immunoglobulin G (IgG) and its concentration is observed in human serum or plasma. RF value higher than 20 international units per milliliter (IU/mL) is considered positive.
Time Frame: Week 24 of the initial treatment, 24 weeks after first re-treatment, and 24 weeks after second retreatment
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 69 | 71
percentage of participants
  Negative: Initial treatment, Week 24 (n=69,71) | 33.3 (273.09) | 38.0 (408.24)
  Positive: Initial treatment, Week 24 (n=69,71) | 66.7 (114.63) | 62.0 (386.02)
  Negative: 1st Retreatment, Week 24 (n=44,43) | 36.4 (79.14) | 48.8 (65.29)
  Positive: 1st Retreatment, Week 24 (n=44,43) | 63.6 (75.68) | 51.2 (41.01)
  Negative: 2nd retreatment, Week 24 (n=15,12) | 46.7 | 83.3
  Positive: 2nd retreatment, Week 24 (n=15,12) | 53.3 | 16.7

18. Secondary Outcome: Percentage of Participants With Anti-cyclic Citrullinated Protein (Anti-CCP) Antibodies at 24 Weeks After Treatment
Description: Anti-CCP antibodies are auto antibodies (antibodies directed against 1 or more of an individual's own proteins) that are frequently detected in the blood of rheumatoid arthritis participants. Anti-CCP antibodies value higher than 10 U/mL is considered positive.
Time Frame: Week 24 of the initial treatment, 24 weeks after first re-treatment, and 24 weeks after second retreatment
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 69 | 71
percentage of participants
  Negative: Initial treatment, Week 24 (n=69,71) | 17.4 | 22.5
  Positive: Initial treatment, Week 24 (n=69,71) | 82.6 | 77.5
  Negative: 1st Retreatment, Week 24 (n=44,43) | 22.7 | 20.9
  Positive: 1st Retreatment, Week 24 (n=44,43) | 77.3 | 79.1
  Negative: 2nd retreatment, Week 24 (n=15,12) | 13.3 | 41.7
  Positive: 2nd retreatment, Week 24 (n=15,12) | 86.7 | 58.3

19. Secondary Outcome: Physician's Global Assessment of Disease Activity
Description: The Physician's Global Assessment of disease activity is assessed on a 0 to 100 millimeter (mm) horizontal VAS by the physician. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm as "maximum disease activity" (maximum arthritis disease activity). Physicians were asked to mark the line and the distance from the left edge was measured. Higher values correspond to worst state of participant (high disease activity).
Time Frame: Day 1 and Week 24 of initial treatment, before 1st retreatment, at 1st retreatment, and at 12 and 24 weeks after 1st retreatment
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 70 | 73
mm
  Initial treatment, Day 1 (n=70,73) | 65.0 (15.0) | 64.1 (15.0)
  Initial treatment, Week 24 (n=69,71) | 27.9 (18.6) | 27.2 (16.2)
  Before 1st retreatment (n=64,63) | 33.7 (17.4) | 26.9 (17.1)
  1st retreatment, Day 1 (n=60,61) | 44.4 (20.8) | 43.3 (18.5)
  1st retreatment, Week 12 (n=56,62) | 30.4 (18.8) | 28.4 (18.0)
  1st retreatment, Week 24 (n=60,59) | 31.9 (19.1) | 24.8 (16.3)

20. Secondary Outcome: Patient Global Assessment of Disease Activity
Description: The Patient's Global Assessment of Disease Activity is assessed on a 0 to 100 mm horizontal VAS by the participant. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm as "maximum disease activity" (maximum arthritis disease activity). Higher values correspond to worst state of participant (high disease activity).
Time Frame: as for outcome 19
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Randomized Re-treatment Arm A: Single 1000 mg IV Rituximab: Participants received rituximab 1000 mg IV on Days 1 and 15. After Week 24, if DAS28 was >3.2, participants received one additional infusion of rituximab 1000 mg IV. Participants received methylprednisolone 100 mg IV 30 minutes before each rituximab infusion and MTX ≥10 mg/week by mouth or parenteral throughout course of treatment.
Arm/Group | Randomized Re-treatment Arm A: Single 1000 mg IV Rituximab | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 70 | 73
mm
  Initial treatment, Day 1 (n=70,73) | 63.0 (20.4) | 64.2 (18.0)
  Initial treatment, Week 24 (n=70,73) | 29.9 (22.3) | 32.6 (22.7)
  Before 1st retreatment (n=65,67) | 33.2 (19.6) | 34.7 (22.3)
  1st retreatment, Day 1 (n=65,66) | 43.7 (21.2) | 46.6 (21.3)
  1st retreatment, Week 12 (n=63,65) | 34.8 (21.2) | 34.5 (25.3)
  1st retreatment, Week 24 (n=64,60) | 35.1 (24.6) | 34.1 (23.1)

21. Secondary Outcome: Patient's Global Assessment of Pain
Description: The participants assessed their pain over the past 24 hours on a 0 to 100 mm horizontal VAS. The left-hand extreme of the line equals 0 mm, and is described as "no pain" and the right-hand extreme equals 100 mm as "unbearable pain". Participants were asked to mark the line and the distance from the left edge was measured. Higher values correspond to worst state of participant (high pain levels).
Time Frame: as for outcome 19
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 70 | 73
mm
  Initial Treatment, Day 1 (n=70,73) | 61.9 (22.3) | 60.1 (19.9)
  Initial Treatment, Week 24 (n=70,73) | 28.5 (22.0) | 30.0 (21.7)
  Before 1st retreatment (n=65,67) | 34.4 (21.3) | 32.9 (23.0)
  1st re-treatment, Day 1 (n=65,67) | 41.1 (21.5) | 45.2 (22.4)
  1st retreatment, Week 12 (n=64,60) | 34.3 (21.4) | 33.9 (25.6)
  1st retreatment, Week 24 (n=64,60) | 34.4 (24.6) | 34.3 (23.7)

22. Secondary Outcome: Participant Assessment of Fatigue
Description: Participants were asked to rate their level of fatigue over the last 7 days on a 100-mm VAS. The left-hand extreme of the line equals 0 mm, and is described as "no fatigue" and the right-hand extreme equals 100 mm as "extreme fatigue". Participants were asked to mark the line and the distance from the left edge was measured. Higher values correspond to worst state of participant (high levels of fatigue).
Time Frame: as for outcome 19
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 70 | 73
mm
  Initial Treatment, Day 1 (n=70,73) | 62.1 (21.4) | 62.0 (22.5)
  Initial Treatment, Week 24 (n=70,73) | 37.1 (24.2) | 39.8 (25.8)
  Before 1st retreatment (n=64,66) | 44.5 (20.8) | 41.2 (26.1)
  1st retreatment, Day 1 (n=65,64) | 50.6 (22.6) | 51.7 (21.6)
  1st retreatment, Week 12 (n=63,65) | 45.2 (23.0) | 45.3 (25.5)
  1st retreatment, Week 24 (n=64,60) | 43.0 (25.3) | 38.9 (23.6)

23. Secondary Outcome: Cortisone Intake AUC (Time- and Weight-Weighted)
Description: All cortisone intakes (in mg) were taken into account (oral, IV [including the cortisone administration before the rituximab infusion], intramuscular, and intra-articular).
Time Frame: Day 1 (each infusion), Week 24, Week 104
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Error); unit: mg*week
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 69 | 73
mg*week
  Day 1 to Week 104 (n=69,73) | 0.08 (0.06) | 0.09 (0.06)
  1st retreatment to Week 104 (n=65,68) | 0.08 (0.06) | 0.09 (0.06)
  Week 24 to Week 104 (n=69,73) | 0.08 (0.06) | 0.09 (0.06)
Statistical Analysis 1: Comparison: Randomized Retreatment Arm A: Rituximab 1000 mg vs Randomized Retreatment Arm B: Rituximab 1000 mg x 2; Day 1 to Week 104; Test type: Superiority or Other; p = 0.389, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Randomized Retreatment Arm A: Rituximab 1000 mg vs Randomized Retreatment Arm B: Rituximab 1000 mg x 2; 1st retreatment to Week 104; Test type: Superiority or Other; p = 0.374, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Randomized Retreatment Arm A: Rituximab 1000 mg vs Randomized Retreatment Arm B: Rituximab 1000 mg x 2; Weel 24 to Week 104; Test type: Superiority or Other; p = 0.277, Wilcoxon (Mann-Whitney)

24. Secondary Outcome: Total Mean Dose of Cortisone Between Week 24 and Week 104
Description: All cortisone intakes were taken into account, including oral, IV (including the cortisone administration before the rituximab infusion), intramuscular and intra-articular.
Time Frame: Week 24 to Week 104
Population: ITT population
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 70 | 73
mg
  Total cortisone: Week 24 to Week 104 | 2542.9 (2085.6) | 2842.5 (2124.9)
  Oral cortisone: Week 24 to Week 104 | 2384.0 (2092.6) | 2425.1 (2046.6)
  IV cortisone: Week 24 to Week 104 | 199.1 (92.3) | 384.9 (193.5)
Statistical Analysis 1: Comparison: Randomized Retreatment Arm A: Rituximab 1000 mg vs Randomized Retreatment Arm B: Rituximab 1000 mg x 2; Total cortisone: Week 24 to Week 104; Test type: Superiority or Other; p = 0.278, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Randomized Retreatment Arm A: Rituximab 1000 mg vs Randomized Retreatment Arm B: Rituximab 1000 mg x 2; Oral cortisone: Week 24 to Week 104; Test type: Superiority or Other; p = 0.887, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Randomized Retreatment Arm A: Rituximab 1000 mg vs Randomized Retreatment Arm B: Rituximab 1000 mg x 2; IV cortisone: Week 24 to Week 104; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

25. Secondary Outcome: HAQ-DI Scores
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0=least difficulty and 3 extreme difficulty.
Time Frame: as for outcome 19
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 70 | 72
units on a scale
  Initial treatment, Day 1 (n=70,69) | 1.74 (0.61) | 1.75 (0.69)
  Initial treatment, Week 24 (n=68,72) | 1.25 (0.67) | 1.31 (0.74)
  Before 1st retreatment (n=64,67) | 1.26 (0.67) | 1.35 (0.73)
  1st retreatment, Day 1 (n=58,58) | 1.32 (0.68) | 1.42 (0.73)
  1st retreatment, Week 12 (n=62,61) | 1.31 (0.66) | 1.33 (0.72)
  1st retreatment, Week 24 (n=63,59) | 1.26 (0.72) | 1.32 (0.72)

26. Secondary Outcome: Short Form 12 (SF-12) Physical Health Composite Score
Description: Physical and Mental Health Composite Scores of SF-12 were computed using the scores of 12 questions and range from 0 to 100, where a 0 score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: as for outcome 19
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 63 | 68
units on a scale
  Initial treatment, Day 1 (n=62,65) | 31.11 (7.55) | 31.07 (7.41)
  Initial Tteatment, Week 24 (n=63,68) | 38.81 (8.39) | 40.05 (8.64)
  Before 1st retreatment (n=21,22) | 39.44 (8.45) | 39.52 (9.99)
  1st retreatment, Day 1 (n=47,44) | 36.57 (6.75) | 35.81 (8.97)
  1st retreatment, Week 12 (n=13,10) | 38.36 (9.30) | 38.05 (10.77)
  1st retreatment, Week 24 (n=40,36) | 36.53 (7.75) | 36.86 (8.13)

27. Secondary Outcome: SF-12 Mental Health Composite Score
Description: Mental Health Composite Scores of SF-12 were computed using the scores of 12 questions and range from 0 to 100, where a 0 score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: as for outcome 19
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 63 | 68
units on a scale
  Initial treatment, Day 1 (n=62,65) | 36.03 (10.03) | 37.13 (9.40)
  Initial treatment, Week 24 (n=63,68) | 43.08 (9.74) | 40.99 (9.01)
  Before 1st retreatment (n=21,22) | 44.94 (9.94) | 41.57 (8.66)
  1st retreatment, Day 1 (n=47,44) | 40.87 (10.53) | 38.52 (7.87)
  1st retreatment, Week 12 (n=13,10) | 41.84 (11.36) | 34.69 (11.06)
  1st retreatment, Week 24 (n=40,36) | 40.90 (10.61) | 41.60 (8.87)

28. Secondary Outcome: Medical Outcomes Study Sleep Scale (MOS-Sleep) Composite Sleep Problems 6 (SLP6) Index
Description: The MOS Sleep Scale measures most constructs of sleep. The scale has a battery of questions to measure specific aspects of sleep in participants with co-morbidities. The SLP6 index is comprised of 6 items: provides a summary of sleep problems and contains questions from the sleep disturbance, sleep adequacy, respiratory impairment, and somnolence domains. The SLP6 index score ranges between 0 and 100, with higher values corresponding to more sleep problems.
Time Frame: as for outcome 19
Population: ITT population;n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 68 | 70
units on a scale
  Initial treatment, Day 1 (n=68,66) | 52.15 (15.32) | 49.89 (15.81)
  Initial treatment, Week 24 (n=65,70) | 43.73 (14.90) | 40.50 (17.17)
  Before 1st retreatment (n=62,65) | 45.44 (13.97) | 41.27 (17.01)
  1st retreatment, Day 1 (n=57,56) | 46.25 (16.53) | 44.94 (16.02)
  1st retreatment, Week 12 (n=61,59) | 43.64 (14.41) | 43.74 (18.60)
  1st retreatment, Week 24 (n=63,59) | 44.74 (15.35) | 40.08 (16.76)

29. Secondary Outcome: Percentage of Participants Reporting Acceptable Disease Activity Symptom State Assessed Using Patient Acceptable and Unacceptable Symptom State (PASS)
Description: Percentage of participants reporting acceptable symptom state: acceptance to remain for the rest of their lives with the level of disease activity they had during the last 48 hours; and unacceptable symptom state: not able to remain for the rest of their lives with the level of disease activity they had during the last 48 hours. In the case of missing data, participants who withdrew from the study because of inefficacy or toxicity were considered "unacceptable".
Time Frame: Week 24, 12 and 24 weeks after 1st retreatment
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 70 | 73
percentage of participants
  Week 24 | 73.4 | 75.4
  1st retreatment, Week 12 | 73.3 | 62.5
  1st retreatment, Week 24 | 70.5 | 64.3

30. Secondary Outcome: Patient Global Assessment of Disease Activity in Participants Reporting Acceptable Symptoms Using PASS
Description: The Patient's Global Assessment of Disease Activity assessed in participants reporting acceptable symptom state using PASS (acceptance to remain for the rest of their lives with the level of disease activity they had during the last 48 hours) on a 0 to 100 mm horizontal VAS by the participant. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm as "maximum disease activity" (maximum arthritis disease activity). Higher values correspond to worst state of participant (high disease activity).
Time Frame: Week 24, 12 and 24 weeks after 1st retreatment
Population: ITT population; only participants with 'acceptable' symptom state assessed using PASS were included in the analysis. n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 47 | 52
mm
  Week 24 (n=47,52) | 23.4 (18.5) | 28.4 (19.1)
  1st retreatment, Week 12 (n=44,35) | 27.4 (16.6) | 27.3 (21.8)
  1st retreatment, Week 24 (n=43,36) | 26.3 (19.5) | 25.7 (16.4)

31. Secondary Outcome: Percentage of Participants With Minimum Clinically Important Improvement (MCII) in Disease Activity
Description: Participants were asked how their disease activity had been during the last 48 hours compared to baseline. Those participants that reported improvement assessed how important this improvement was to them; range: very important, moderately important, slightly important, or not at all important. Binary response options: 1=improved very important, or improved moderately important; 2=slightly important, not at all important, no change, or worse-more disease activity.
Time Frame: Week 24, 12 and 24 weeks after 1st retreatment
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 70 | 73
percentage of participants
  Week 24 | 75.4 | 81.2
  1st retreatment, Week 12 | 65.6 | 63.0
  1st retreatment, Week 24 | 66.7 | 66.1

32. Secondary Outcome: Change From Baseline in Patient Global Assessment of Disease Activity in Participants With MCII
Description: The Patient's Global Assessment of Disease Activity was assessed in participants reporting MCII on a 0 to 100 mm horizontal VAS by the participant. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm as "maximum disease activity" (maximum arthritis disease activity). Higher values correspond to worst state of participant (high disease activity).
Time Frame: Baseline, Week 24, 12 and 24 weeks after 1st retreatment
Population: ITT population; only participants with MCII were included in the analysis. n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 49 | 56
mm
  Week 24 (n=49,56) | -12.4 (20.7) | -4.6 (22.9)
  1st retreatment, Week 12 (n=38,30) | -4.2 (16.0) | -9.2 (17.7)
  1st retreatment, Week 24 (n=40,37) | -2.5 (17.8) | -2.9 (20.6)

33. Secondary Outcome: Percentage of Participants Reporting Acceptable Symptom State in Functioning Assessed Using PASS
Description: Percentage of participants reporting acceptable symptom state: acceptance to remain for the rest of their lives with the level of function they had during the last 48 hours; and unacceptable symptom state: not able to remain for the rest of their lives with the level of function they had during the last 48 hours. In the case of missing data, participants who withdrew from the study because of inefficacy or toxicity were considered "unacceptable".
Time Frame: Week 24, 12 and 24 weeks after 1st retreatment
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 70 | 73
percentage of participants
  Week 24 | 74.2 | 72.7
  1st retreatment, Week 12 | 75.9 | 60.0
  1st retreatment, Week 24 | 70.2 | 62.1

34. Secondary Outcome: HAQ-DI Scores in Participants Reporting Acceptable Function Using PASS
Description: HAQ-DI was assessed in participants reporting acceptable symptom state using PASS (acceptance to remain for the rest of their lives with the level of disease activity they had during the last 48 hours). HAQ-DI is a participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0=least difficulty and 3 extreme difficulty.
Time Frame: Week 24, 12 and 24 weeks after 1st retreatment
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 46 | 48
units on a scale
  Week 24 (n=46,48) | 1.16 (0.69) | 1.16 (0.74)
  1st retreatment, Week 12 (n=44,33) | 1.20 (0.70) | 1.08 (0.71)
  1st retreatment, Week 24 (n=40,36) | 1.14 (0.75) | 1.08 (0.72)

35. Secondary Outcome: Percentage of Participants With MCII in Functioning
Description: Participants were asked how their functioning had been during the last 48 hours compared to baseline. Those participants that reported improvement assessed how important this improvement was to them; range: very important, moderately important, slightly important, or not at all important. Binary response options: 1=improved very important, or improved moderately important; 2=slightly important, not at all important, no change, or worse.
Time Frame: Week 24, 12 and 24 weeks after 1st retreatment
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 70 | 73
percentage of participants
  Week 24 | 73.4 | 76.5
  1st retreatment, Week 12 | 65.0 | 63.0
  1st retreatment, Week 24 | 65.5 | 57.9

36. Secondary Outcome: Change From Baseline in HAQ-DI in Participants With MCII
Description: HAQ-DI was assessed in participants with MCII. HAQ-DI is a participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0=least difficulty and 3 extreme difficulty.
Time Frame: Baseline, Week 24, 12 and 24 weeks after 1st retreatment
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 47 | 52
units on a scale
  Week 24 (n=47,52) | -0.11 (0.46) | -0.06 (0.56)
  1st retreatment, Week 12 (n=38,30) | -0.03 (0.30) | -0.11 (0.39)
  1st retreatment, Week 24 (n=38,30) | -0.07 (0.24) | -0.09 (0.29)

37. Secondary Outcome: Percentage of Participants With Acceptable Symptom State in Pain Assessed Using PASS
Description: Percentage of participants reporting acceptable symptom state: acceptance to remain for the rest of their lives with the level of pain they had during the last 48 hours; and unacceptable symptom state: not able to remain for the rest of their lives with the level of pain they had during the last 48 hours. In the case of missing data, participants who withdrew from the study because of inefficacy or toxicity were considered "unacceptable".
Time Frame: Week 24, 12 and 24 weeks after 1st retreatment
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 70 | 73
percentage of participants
  Week 24 | 74.2 | 75.0
  1st retreatment Week 12 | 70.2 | 61.8
  1st retreatment, Week 24 | 72.9 | 61.4

38. Secondary Outcome: Patient Global Assessment of Pain in Participants Reporting Acceptable Symptoms Using PASS
Description: Patient Global Assessment of Pain assessed in participants reporting acceptable symptom state using PASS (acceptance to remain for the rest of their lives with the level of pain they had during the last 48 hours) on a 0 to 100 mm horizontal VAS by the participant. The left-hand extreme of the line equals 0 mm, and is described as "no pain" and the right-hand extreme equals 100 mm as "unbearable pain". Higher values correspond to worst state of participant (high pain levels).
Time Frame: Week 24, 12 and 24 weeks after 1st retreatment
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 46 | 51
mm
  Week 24 (n=46,51) | 21.5 (16.2) | 26.4 (18.5)
  1st retreatment, Week 12 (n=40,34) | 26.8 (17.3) | 27.6 (22.4)
  1st retreatment, Week 24 (n=43,35) | 26.3 (20.1) | 25.1 (17.3)

39. Secondary Outcome: Percentage of Participants With MCII in Pain
Description: Participants were asked how their pain had been during the last 48 hours compared to baseline. Those participants that reported improvement assessed how important this improvement was to them; range: very important, moderately important, slightly important, or not at all important. Binary response options: 1=improved very important, or improved moderately important; 2=slightly important, not at all important, no change, or worse pain.
Time Frame: Week 24, 12 and 24 weeks after 1st retreatment
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 63 | 70
percentage of participants
  Week 24 (n=63,70) | 76.2 | 80.0
  1st retreatment, Week 12 (n=59,55) | 71.2 | 69.1
  1st retreatment, Week 24 (n=61,57) | 68.9 | 61.4

40. Secondary Outcome: Change From Baseline in Patient Global Assessment of Pain in Participants With MCII
Description: as for outcome 21
Time Frame: Baseline, Week 24, 12 and 24 weeks after 1st retreatment
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2
Number analyzed (Participants) | 48 | 56
mm
  Week 24 (n=48,56) | -13.5 (21.0) | -4.3 (23.9)
  1st retreatment, Week 12 (n=39,35) | -2.7 (13.6) | -8.9 (16.4)
  1st retreatment, Week 24 (n=42,35) | -3.5 (24.3) | -3.2 (18.4)

ADVERSE EVENTS:
Time Frame: Baseline to 104 weeks; related serious adverse events (SAEs) were collected and reported regardless of time elapsed from last dose of study drug; unrelated SAEs were collected during the study and for up to 24 weeks after last dose of study drug.
Arm/Group | Randomized Retreatment Arm A: Rituximab 1000 mg | Randomized Retreatment Arm B: Rituximab 1000 mg x 2 | Nonrandomized: Rituximab 1000 mg
Serious Adverse Events (participants affected / at risk) | 19/66 | 25/68 | 16/81
Other Adverse Events (participants affected / at risk) | 61/66 | 65/68 | 72/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Retreatment Arm A: Rituximab 1000 mg (N=66) | Randomized Retreatment Arm B: Rituximab 1000 mg x 2 (N=68) | Nonrandomized: Rituximab 1000 mg (N=81)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 4 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bone erosion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Abdominal wall abscess (Infections and infestations) | 1 | 0 | 0
Bursitis infective (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Hepatitis B (Infections and infestations) | 0 | 1 | 0
Perianal abscess (Infections and infestations) | 1 | 0 | 0
Pertussis (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Prostate infection (Infections and infestations) | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cyst (General disorders) | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1
Mania (Psychiatric disorders) | 0 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 1
Vasculitis (Vascular disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Goitre (Endocrine disorders) | 1 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0 | 0
Bartholinitis (Reproductive system and breast disorders) | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Retreatment Arm A: Rituximab 1000 mg (N=66) | Randomized Retreatment Arm B: Rituximab 1000 mg x 2 (N=68) | Nonrandomized: Rituximab 1000 mg (N=81)
Bronchitis (Infections and infestations) | 13 | 16 | 11
Urinary tract infection (Infections and infestations) | 9 | 12 | 14
Gastroenteritis (Infections and infestations) | 8 | 10 | 3
Nasopharyngitis (Infections and infestations) | 7 | 6 | 2
Rhinitis (Infections and infestations) | 3 | 4 | 6
Pharyngitis (Infections and infestations) | 4 | 6 | 2
Tonsillitis (Infections and infestations) | 4 | 3 | 0
Sinusitis (Infections and infestations) | 4 | 2 | 1
Influenza (Infections and infestations) | 3 | 3 | 0
Oral herpes (Infections and infestations) | 1 | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 3 | 0
Bronchopneumonia (Infections and infestations) | 2 | 1 | 0
Fungal skin infection (Infections and infestations) | 2 | 0 | 1
Localised infection (Infections and infestations) | 0 | 2 | 1
Tracheitis (Infections and infestations) | 2 | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 1 | 0
Fungal infection (Infections and infestations) | 2 | 0 | 0
Onychomycosis (Infections and infestations) | 1 | 0 | 1
Oral fungal infection (Infections and infestations) | 0 | 2 | 0
Rhinotracheitis (Infections and infestations) | 0 | 1 | 1
Sinobronchitis (Infections and infestations) | 1 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 1
Abdominal wall abscess (Infections and infestations) | 1 | 0 | 0
Bronchiectasis (Infections and infestations) | 0 | 1 | 0
Bursitis infective (Infections and infestations) | 1 | 0 | 0
Campylobacter intestinal infection (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Hepatitis B (Infections and infestations) | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0
Infected sebaceous cyst (Infections and infestations) | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0
Perianal abscess (Infections and infestations) | 1 | 0 | 0
Pertussis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Prostate infection (Infections and infestations) | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 1 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1
Vaginal candidiasis (Infections and infestations) | 0 | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 8 | 12 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 10 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 6 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Bone erosion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Toe deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Asthenia (General disorders) | 11 | 11 | 6
Pyrexia (General disorders) | 3 | 4 | 4
Fatigue (General disorders) | 1 | 1 | 3
Oedema peripheral (General disorders) | 1 | 2 | 1
Feeling hot (General disorders) | 2 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 2
Drug intolerance (General disorders) | 0 | 1 | 0
Face oedema (General disorders) | 0 | 1 | 1
Malaise (General disorders) | 0 | 2 | 0
Oedema (General disorders) | 1 | 1 | 0
Adverse drug reaction (General disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 1 | 0 | 0
Chills (General disorders) | 0 | 1 | 0
Cyst (General disorders) | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 1 | 0
Infusion site phlebitis (General disorders) | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 1 | 0
Localised oedema (General disorders) | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Sense of oppression (General disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 5 | 6
Abdominal pain upper (Gastrointestinal disorders) | 5 | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 2
Vomiting (Gastrointestinal disorders) | 4 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 3 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 2 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 2 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 7 | 11 | 10
Sciatica (Nervous system disorders) | 3 | 6 | 4
Migraine (Nervous system disorders) | 0 | 3 | 1
Restless legs syndrome (Nervous system disorders) | 1 | 1 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0
Cervical root pain (Nervous system disorders) | 1 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 1
Dystonia (Nervous system disorders) | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Parkinsonism (Nervous system disorders) | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 4 | 3
Larynx irritation (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 6 | 5
Rash (Skin and subcutaneous tissue disorders) | 4 | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 3 | 2
Eczema (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema nummular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 2 | 0
Limb injury (Injury, poisoning and procedural complications) | 2 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Stress fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7 | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetes mellitus non-insulin-dependent (Metabolism and nutrition disorders) | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 4 | 1 | 3
Hot flush (Vascular disorders) | 3 | 2 | 3
Hypertensive crisis (Vascular disorders) | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 2
Arteriosclerosis (Vascular disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 1 | 0
Vasculitis (Vascular disorders) | 1 | 0 | 0
Venous insufficiency (Vascular disorders) | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 2 | 5 | 5
Insomnia (Psychiatric disorders) | 0 | 4 | 2
Anxiety (Psychiatric disorders) | 1 | 3 | 0
Sleep disorder (Psychiatric disorders) | 2 | 1 | 0
Depressive symptom (Psychiatric disorders) | 0 | 1 | 0
Mania (Psychiatric disorders) | 0 | 0 | 1
Transaminases increased (Investigations) | 2 | 1 | 1
Weight increased (Investigations) | 2 | 1 | 1
Eosinophil count increased (Investigations) | 1 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 1
Hepatic enzyme increased (Investigations) | 0 | 2 | 0
Weight decreased (Investigations) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Bacteria urine identified (Investigations) | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0
Blood phosphorus decreased (Investigations) | 1 | 0 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0 | 0
Cardiac murmur (Investigations) | 0 | 1 | 0
Deoxyribonucleic acid (DNA) antibody positive (Investigations) | 1 | 0 | 0
Electrocardiogram repolarisation abnormality (Investigations) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0
Neutrophil count increased (Investigations) | 1 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 5 | 1 | 0
Cataract (Eye disorders) | 1 | 1 | 1
Dry eye (Eye disorders) | 2 | 0 | 1
Chalazion (Eye disorders) | 1 | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 1
Visual disturbance (Eye disorders) | 0 | 0 | 2
Eye irritation (Eye disorders) | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0
Keratitis (Eye disorders) | 0 | 1 | 0
Keratoconjunctivitis sicca (Eye disorders) | 1 | 0 | 0
Ocular discomfort (Eye disorders) | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1
Ocular hypertension (Eye disorders) | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1
Retinopathy hypertensive (Eye disorders) | 1 | 0 | 0
Uveitis (Eye disorders) | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 2 | 3
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocythaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 5 | 1 | 3
Tinnitus (Ear and labyrinth disorders) | 1 | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Vaginal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 3 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Bundle branch block left (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 3 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Hypertonic bladder (Renal and urinary disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Bartholinitis (Reproductive system and breast disorders) | 0 | 2 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Cataract operation (Surgical and medical procedures) | 1 | 1 | 1
Apicectomy (Surgical and medical procedures) | 0 | 1 | 0
Corneal operation (Surgical and medical procedures) | 0 | 1 | 0
Skin neoplasm excision (Surgical and medical procedures) | 1 | 0 | 0
Therapy regimen changed (Surgical and medical procedures) | 0 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 1 | 0
Cytolytic hepatitis (Hepatobiliary disorders) | 0 | 2 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 2
Allergy to chemicals (Immune system disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
Goitre (Endocrine disorders) | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Nonserious adverse events (AEs) presented in this record include all AEs reported during the study, not just nonserious events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.